CLINICAL TRIAL: NCT02033044
Title: Randomized Controlled Trial Comparing the Effects on Psychosocial Functioning of Cognitive Rehabilitation Versus Psychoeducation in Borderline Personality Disorder
Brief Title: Cognitive Rehabilitation Versus Psychoeducation in Psychosocial Functioning of Borderline Personality Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Jose Luis Carrasco, Head Professor Department of Psychiatry, MD., Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COGREHAB
Record Dates: First submitted 2013-12-23; First posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Neuropsychology
Keywords: borderline personality disorder; cognitive rehabilitation; psychoeducation; psychosocial functioning
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Cognitive Remediation; Cognitive Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cognitive remediation (Experimental): Cognitive remediation programme in order to improve several cognitive domains.
  Interventions: Other: cognitive remediation
- Psychoeducation (Active Comparator): Psychoeducation group in order to improve psychosocial functioning of patients.
  Interventions: Other: Psychoeducation

INTERVENTIONS:
Other: cognitive remediation — Cognitive Rehabilitation (CR). Consisted on group sessions (5 individuals per group) of 120-minutes, twice a week during a total period of 16 weeks (32 sessions). The exercises addressed neurocognitive issues related to sustained attention, processing speed, memory and executive functioning. The whole program aimed at getting new strategies to improve functional adaptation, thus tasks were carried out in the clinical setting and at home. Some homework tasks were based on their daily life difficulties and problems. The main objective of this program was the generalization of rehabilitated cognitive functions to daily life activities. Most of the techniques were based on a previous program for bipolar disorder.
  Other Names: Cognitive rehabilitation
  Arms: cognitive remediation
Other: Psychoeducation — Psychoeducation (PE). The psychoeducation intervention consisted of 16 weekly group sessions of 5 individuals of 120 minutes each (16 sessions). This therapy aimed at improving illness' consciousness , interpersonal abilities, family balance, therapeutical adherence, emotional management in frustrating situations, problems resolutions, and lifestyle regularity. On this intervention, no homework tasks were required. This intervention was based on the Systems Training for Emotional Predictability and Problem Solving (STEPPS) program therapy.
  Other Names: Psychoeducation Programme
  Arms: Psychoeducation

SUMMARY:
Study design was a multicenter, randomized, rater-blind clinical trial. There were two-parallel arms (1:1) to evaluate functional, clinical and cognitive efficacy of a specific cognitive rehabilitation group intervention (CR) compared with a psychoeducational group intervention (PE) in subjects with Borderline Personality Disorder (BPD).

DETAILED DESCRIPTION:
To ensure the reliability among centers regarding the evaluation and the treatment fidelity, two meetings were organized before the start of the study to train therapists in the evaluations and interventions.

Clinical and neuropsychological evaluations before interventions were administered in different days since they lasted in general more than one hour each one and the effect of fatigue or boredom might affect the results. Clinical interviews were performed by experienced psychiatrists and psychologists during 3 months to ensure the follow-up of all participants prospectively. The following sociodemographic and clinical variables were collected: age at recruitment, gender, education level, occupational status, and pharmacological treatment. All participants were then randomized to receive CR or PE in a 1:1 ratio stratified by center, age, and education level. Randomization was accomplished with the use of computer-generated sequence.

During the study, subjects did not receive any other individual or group psychotherapy. All patients continued pharmacological treatment if it had been initiated prior to inclusion. Type and doses of medication could not be modified during the study period. Both interventions were applied in a group format and were conducted by two psychologists with experience in managing patients with BPD. Subjects were instructed not to disclose any information about the intervention to maintain blind conditions. Participants were evaluated at baseline, after completion of the intervention, and six months after the end of the interventions.

The study was conducted in accordance with the ethical principles of the Declaration of Helsinki and the approval of the Ethical Committee for this study was obtained. All subjects received extensive information about the study and provided written informed consent before they were enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients aged 18 to 45 years;
* Diagnoses of BPD according to Diagnostic and Statistical Manual for Mental Disorders (4th version Revised) (DSM-IV-TR) criteria and evaluated by two semi-structured diagnostic interviews
* Structured Clinical Interview for DSM-IV Axis II Disorders (SCID-II) and the Revised Diagnostic Interview for Borderlines (DIB-R)
* Clinical severity measured with Clinical Global Impression for BPD (CGI-BPD) higher than 4;
* Functional impairment measured with a Global Assessment Functioning (GAF) lower than 65.

Exclusion Criteria:

* No severe physical conditions, such as organic brain syndrome or neurological disease that could affect neuropsychological performance;
* Intelligence Quotient (IQ) < 85;
* Major Depression Disorder (MDD) or substance misuse within the last 6 months;
* Schizophrenia, severe psychotic disorder or bipolar disorder;
* Previous participation in any psychoeducation or cognitive rehabilitation intervention.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2010-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Functioning Assessment Scale Test (FAST) | up to three years
  This test is a 24-item scale that measures the level of psychosocial functioning of patients in daily life situations. It assesses six functional domains: autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal relationships, and leisure time. Higher scores indicate higher functional impairment. This instrument has shown good psychometric properties and sensitivity to change.

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Carrasco, MD, Principal Investigator — Hospital Clinico San Carlos; Juan C Pascual, MD, Study Chair — Hospital San Creu i San Pau; Angela Ibañez, MD, Study Chair — Hospital Universitario Ramon y Cajal
Locations (1):
- Hospital Clinico San Carlos, Madrid, Madrid, Spain

REFERENCES:
- [Background] Torrent C, Bonnin Cdel M, Martinez-Aran A, Valle J, Amann BL, Gonzalez-Pinto A, Crespo JM, Ibanez A, Garcia-Portilla MP, Tabares-Seisdedos R, Arango C, Colom F, Sole B, Pacchiarotti I, Rosa AR, Ayuso-Mateos JL, Anaya C, Fernandez P, Landin-Romero R, Alonso-Lana S, Ortiz-Gil J, Segura B, Barbeito S, Vega P, Fernandez M, Ugarte A, Subira M, Cerrillo E, Custal N, Menchon JM, Saiz-Ruiz J, Rodao JM, Isella S, Alegria A, Al-Halabi S, Bobes J, Galvan G, Saiz PA, Balanza-Martinez V, Selva G, Fuentes-Dura I, Correa P, Mayoral M, Chiclana G, Merchan-Naranjo J, Rapado-Castro M, Salamero M, Vieta E. Efficacy of functional remediation in bipolar disorder: a multicenter randomized controlled study. Am J Psychiatry. 2013 Aug;170(8):852-9. doi: 10.1176/appi.ajp.2012.12070971. PMID 23511717
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Pascual JC, Palomares N, Ibanez A, Portella MJ, Arza R, Reyes R, Feliu-Soler A, Diaz-Marsa M, Saiz-Ruiz J, Soler J, Carrasco JL. Efficacy of cognitive rehabilitation on psychosocial functioning in Borderline Personality Disorder: a randomized controlled trial. BMC Psychiatry. 2015 Oct 21;15:255. doi: 10.1186/s12888-015-0640-5. PMID 26487284